CLINICAL TRIAL: NCT04018027
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Oral Difelikefalin (CR845) for Moderate to Severe Pruritus in Adult Subjects With Atopic Dermatitis
Brief Title: Study to Evaluate the Efficacy and Safety of Oral Difelikefalin (CR845) for Moderate to Severe Pruritus in Subjects With Atopic Dermatitis
Acronym: KARE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cara Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR845-210501
Record Dates: First submitted 2019-07-09; First posted 2019-07-12 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Pruritus; Atopic Dermatitis
Keywords: Atopic Dermatitis; Pruritus; CR845; Chronic Itch; difelikefalin; Itch; Itching; Generalized pruritus; Eczema
MeSH Terms: conditions — Pruritus; Dermatitis, Atopic; Eczema | interventions — difelikefalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Difelikefalin 0.25 mg (Active Comparator): Oral difelikefalin 0.25 mg tablet administered twice daily
  Interventions: Drug: difelikefalin 0.25 mg
- Difelikefalin 0.5 mg (Active Comparator): Oral difelikefalin 0.5 mg tablet administered twice daily
  Interventions: Drug: difelikefalin 0.5 mg
- Difelikefalin 1.0 mg (Active Comparator): Oral difelikefalin 1.0 mg tablet administered twice daily
  Interventions: Drug: difelikefalin 1.0 mg
- Placebo (Placebo Comparator): Oral placebo tablet administered twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: difelikefalin 0.25 mg — Oral difelikefalin 0.25 mg administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 0.25 mg
Drug: difelikefalin 0.5 mg — Oral difelikefalin 0.5 mg administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 0.5 mg
Drug: difelikefalin 1.0 mg — Oral difelikefalin 1.0 mg administered twice daily
  Other Names: CR845
  Arms: Difelikefalin 1.0 mg
Drug: Placebo — Oral Placebo administered twice daily
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, 4-arm, placebo-controlled study to evaluate the efficacy and safety of twice-daily (BID) oral difelikefalin (CR845) in adult subjects with atopic dermatitis (AD) and moderate to severe pruritus.

DETAILED DESCRIPTION:
The study will consist of a 30-day Screening period, a 7-day Run-In period, a 12-week Placebo-Controlled Treatment period followed by a 4-week Active Extension period and a Follow Up visit approximately 7 days after the last dose of study drug.

All subjects will sign an informed consent form (ICF) and undergo screening for study eligibility.

Subjects will be randomized to receive either placebo or difelikefalin (CR845) tablets at a dose of 0.25 mg, 0.5 mg, or 1.0 mg, orally BID. Intake of the first dose of study drug will be at Day 1.

Subjects who complete the Placebo-Controlled Treatment period of the study will transition into the Active Extension upon completion of the Week 12 visit assessments. All subjects in the Active Extension will receive difelikefalin (CR845).

ELIGIBILITY:
Key Inclusion Criteria:

To be eligible for inclusion into the study, a patient must meet the following criteria:

* Subject has clinically confirmed diagnosis of active AD;
* Subject has at least a 12-month history of AD;
* Subject has chronic itch related to AD;
* Subject has moderate to severe pruritus;
* Female subject is not pregnant or nursing during any period of the study.

Key Exclusion Criteria:

A patient will be excluded from the study if any of the following criteria are met:

* Subject has clinically infected AD;
* Subject has pruritus attributed to a cause other than AD;
* Subject has any clinically significant medical condition or physical/laboratory/ECG/vital signs abnormality that would, in the opinion of the investigator, put the subject at undue risk or interfere with interpretation of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2019-06-29 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the weekly mean of the daily 24-hour Itch-Numeric Rating Scale (I-NRS) score at Week 12. | Baseline, Week 12

SECONDARY OUTCOMES:
Reduction of itch intensity as assessed by the proportion of patients achieving an improvement from baseline ≥4 points with respect to the weekly mean of the daily 24-hour I-NRS score at Week 12 | Week 12
Improvement in itch-related quality of life as assessed by the change from baseline to Week 12 in 5-D Itch Scale score | Baseline, Week 12
Improvement in itch-related quality of life as assessed by the change from baseline to Week 12 in total Skindex-10 Scale score | Baseline, Week 12
Improvement in itch-related quality of life as assessed by the change from baseline to Week 12 in Sleep Quality Assessment. | Baseline, Week 12
Percent of subjects with adverse events. | Baseline, Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Kristine Nograles, Study Director — Cara Therapeutics
Locations (39):
- United States (37):
  - Cara Therapeutics Study Site, Anniston, Alabama
  - Cara Therapeutics Study Site, Birmingham, Alabama
  - Cara Therapeutics Study Site, Scottsdale, Arizona
  - Cara Therapeutics Study Site, Bryant, Arkansas
  - Cara Therapeutics Study Site, Fountain Valley, California
  - Cara Therapeutics Study Site, Lomita, California
  - Cara Therapeutics Study Site, Cromwell, Connecticut
  - Cara Therapeutics Study Site, Farmington, Connecticut
  - Cara Therapeutics Study Site, Aventura, Florida
  - Cara Therapeutics Study Site 2, Miami, Florida
  - Cara Therapeutics Study Site, Miami, Florida
  - Cara Therapeutics Study Site, Miami Lakes, Florida
  - Cara Therapeutics Study Site, Ocala, Florida
  - Cara Therapeutics Study Site, Sarasota, Florida
  - Cara Therapeutics Study Site, Sweetwater, Florida
  - Cara Therapeutics Study Site, Columbus, Georgia
  - Cara Therapeutics Study Site, Boise, Idaho
  - Cara Therapeutics Study Site 2, Boise, Idaho
  - Cara Therapeutics Study Site, Baton Rouge, Louisiana
  - Cara Therapeutics Study Site, Metairie, Louisiana
  - Cara Therapeutics Study Site, New Orleans, Louisiana
  - Cara Therapeutics Study Site, Brighton, Massachusetts
  - Cara Therapeutics Study Site 2, Las Vegas, Nevada
  - Cara Therapeutics Study Site, Berlin, New Jersey
  - Cara Therapeutics Study Site, Horseheads, New York
  - Cara Therapeutics Study Site, New York, New York
  - Cara Therapeutics Study Site, Cleveland, Ohio
  - Cara Therapeutics Study Site, Oklahoma City, Oklahoma
  - Cara Therapeutics Study Site, Tulsa, Oklahoma
  - Cara Therapeutics Study Site, Medford, Oregon
  - Cara Therapeutics Study Site, Rapid City, South Dakota
  - Cara Therapeutics Study Site 2, Austin, Texas
  - Cara Therapeutics Study Site, Austin, Texas
  - Cara Therapeutics Study Site, Cypress, Texas
  - Cara Therapeutics Study Site, Dallas, Texas
  - Cara Therapeutics Study Site, Salt Lake City, Utah
  - Cara Therapeutics Study Site, Richmond, Virginia
- Canada (2):
  - Cara Therapeutics Study Site, London, Ontario
  - Cara Therapeutics Study Site, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No